CLINICAL TRIAL: NCT04042493
Title: Dissemination and Implementation of Effective Childhood Obesity Treatment Innovations
Brief Title: Connect for Health Pediatric Weight Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Denver Health and Hospital Authority (Other); Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P002972; DI-2017C3-9005 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Overweight and Obesity; Severe Obesity
Keywords: Overweight; Obesity; Pediatric; Implementation; Dissemination
MeSH Terms: conditions — Overweight; Obesity; Obesity, Morbid | interventions — Health

STUDY DESIGN:
Intervention Model Description: The Connect for Health program is a package of practice-level care enhancements to systematically improve the quality of clinical care provided for childhood obesity and offer support directly to parents to improve the children's growth trajectories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connect for Health Program (Experimental)
  Interventions: Behavioral: Connect for Health

INTERVENTIONS:
Behavioral: Connect for Health — The program includes (1) electronic health record (EHR)-based clinical decision support tools to guide pediatric providers in child weight management; (2) clinician and medical staff training in obesity management best practices, (3) family educational materials focused on evidence-based behavioral targets; and (4) social- and community-informed text messages for parents to support behavior change.

SUMMARY:
The overall aim of this study is to disseminate the evidence-based Connect for Health program, specifically targeting pediatric primary care practices that deliver care to low-income children in the US who have a disproportionately high prevalence of childhood obesity and evaluate the effectiveness of the program implementation and dissemination.

ELIGIBILITY:
Inclusion Criteria:

* All children receiving primary care at the participating health centers across the three health systems

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19304 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in child Body Mass Index | One year
  Age- and sex-specific Body Mass Index z-score

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Greenville Health System / Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simione M, Aschbrenner K, Farrar-Muir H, Luo M, Granadeno J, Caballero-Gonzalez A, Price SN, Torres C, Boudreau AA, Fiechtner L, Hambidge SJ, Sease K, Taveras EM. Adapting Connect for Health pediatric weight management program for telehealth in response to the COVID-19 pandemic. Implement Sci Commun. 2023 Nov 16;4(1):139. doi: 10.1186/s43058-023-00523-2. PMID 37974245
- [Derived] Simione M, Farrar-Muir H, Mini FN, Perkins ME, Luo M, Frost H, Orav EJ, Metlay J, Zai AH, Kistin CJ, Sease K, Hambidge SJ, Taveras EM; Connect for Health Collaborative. Implementation of the Connect for Health pediatric weight management program: study protocol and baseline characteristics. J Comp Eff Res. 2021 Aug;10(11):881-892. doi: 10.2217/cer-2021-0076. Epub 2021 May 24. PMID 34024120
- [Derived] Simione M, Frost HM, Cournoyer R, Mini FN, Cassidy J, Craddock C, Moreland J, Wallace J, Metlay J, Kistin CJ, Sease K, Hambidge SJ, Taveras EM. Engaging stakeholders in the adaptation of the Connect for Health pediatric weight management program for national implementation. Implement Sci Commun. 2020 Jun 17;1:55. doi: 10.1186/s43058-020-00047-z. eCollection 2020. PMID 32885211